CLINICAL TRIAL: NCT07042464
Title: Effect of Modified Poco-Poco Exercise to Global DNA Methylation, Growth Differentiation Factor-15, and Sarcopenia Staging in Elderly
Brief Title: Effect of Modified Poco-Poco Exercise to Aging Biomarkers in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKFR.11_2.06.25
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Geriatrics Rehabilitation

STUDY DESIGN:
Intervention Model Description: All research subjects received modified poco-poco exercise program for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified poco-poco exercises (Experimental): Participants performed modified poco-poco exercises three times weekly for 12 weeks and were assessed, including sarcopenia staging (determined by assessing skeletal muscle index, muscle strength, physical performance) and levels of global DNA methylation and GDF-15
  Interventions: Procedure: Modified poco-poco exercises

INTERVENTIONS:
Procedure: Modified poco-poco exercises — Participants performed modified poco-poco exercises three times weekly for 12 weeks

SUMMARY:
Subject with sarcopenia get modified poco-poco exercise program for 12 weeks

DETAILED DESCRIPTION:
34 participants (>60 years) with sarcopenia were modified poco-poco exercises three times weekly for 12 weeks will assessed sarcopenia staging (determined by assessing skeletal muscle index, muscle strength, physical performance) and levels of global DNA methylation and GDF-15.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years old
* Have sarcopenia (based on AWGSOP 2019 criteria)

Exclusion Criteria:

* Hearing impairment/loss hindering participants to receive verbal instructions
* Vision impairment/loss hindering participants to receive instructions
* Musculoskeletal impairment or severe joint diseases (i.e. deformity in Osteoarthritis or Rheumatoid Arthritis)
* Participants have been involved in other exercise program
* Severe cardiovascular disease diagnosed by Cardiologist.
* Participants will be excluded from the research if they skip 3 sessions of the program consecutively or skip 5 sessions cumulatively

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia Staging (Skeletal Muscle Index) | 12 weeks
  Skeletal muscle index
Sarcopenia Staging (Muscle Strength) | 12 weeks
  Hand Grip Strength, score in kilograms
Sarcopenia Staging (Physical Performance) | 12 weeks
  Short Physical Performance Battery, score in numerical 0-12
Levels of Global DNA Methylation | 12 weeks
  Global DNA methylation levels were analyzed using the ELISA-based kit
Levels of Growth Differentiation Factor 15 | 12 weeks
  Growth Differentiation Factor 15 were analyzed the Quantikine ELISA Human GDF-15 Immunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Sadikin General Hospital, Bandung, Indonesia